CLINICAL TRIAL: NCT00062881
Title: Phase I Study of Intrathecal Mafosfamide
Brief Title: Intrathecal Mafosfamide
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Susan Blaney, Professor, Pediatrics-Hema & Oncology, Baylor College of Medicine
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H3241; I.T. Mafosfamide
Record Dates: First submitted 2003-06-17; First posted 2003-06-18 (Estimated); Last update posted 2020-03-04 (Actual); Status verified 2020-03

CONDITIONS: Malignant Meningeal Neoplasms
Keywords: Cancer; Leukemia; Lymphoma; Solid Tumor
MeSH Terms: conditions — Meningeal Neoplasms; Neoplasms; Leukemia; Lymphoma

INTERVENTIONS:
Drug: Intrathecal Mafosfamide

SUMMARY:
This research study is an investigational treatment with the experimental drug Mafosfamide. This treatment is only for children with cancer that has spread to the meninges (tissues that cover the spinal column and brain) and has continued to grow despite treatment with standard therapy.

Mafosfamide is a drug reported to have antitumor effects in animals and that has been given safely into the cerebrospinal fluid (the fluid within and surrounding the brain) in a small number of children and adults. Since there is limited experience in adults and children in giving mafosfamide in this way, the main purpose of this study is to determine the appropriate safe dose of mafosfamide when given intrathecally, that is directly into the cerebrospinal fluid.

The purposes for this study are to (a) determine what dose of mafosfamide can be safely given into the cerebrospinal fluid through an Ommaya reservoir (surgically implanted catheters used to sample cerebrospinal fluid and to instill medication into the cerebrospinal fluid) and lumbar puncture (spinal tap) or lumbar reservoir; (b) look for side effects of drug treatment; (c) to study the pharmacology (how the human body handles the drug) when given directly into the spinal fluid; and (d) see if this drug is beneficial to the patient.

DETAILED DESCRIPTION:
Mafosfamide is given directly into the cerebrospinal fluid twice a week for six successive weeks. If after six weeks the disease has not shown any evidence of progression (tumor growth) patients will continue to receive intrathecal (I.T.) mafosfamide once a week for one month, followed by twice monthly (every other week) for four months, followed by once a month. Patients may continue to receive mafosfamide as long as unacceptable side effects do not occur and there is no growth of the tumor.

Patients will have a weekly physical exam and blood tests. The cerebrospinal fluid will be tested each time they receive drug for the presence of cancer cells. If the patient has an Ommaya reservoir (a surgically implanted catheter that is used to sample cerebrospinal fluid from the fluid chambers in the head and to install medication into the cerebrospinal fluid) then the doctor may recommend that they receive one dose of mafosfamide through the Ommaya reservoir and the next dose via lumbar puncture (spinal tap) or lumbar reservoir. A lumbar reservoir is a catheter that is surgically implanted into the lower back. This catheter is used to sample cerebrospinal fluid and to install medication into the cerebrospinal fluid.

All patients must be observed for a minimum of eight hours after the first dose of intrathecal mafosfamide. If the first dose is well tolerated (there are no major side effects), further doses of mafosfamide will be administered with close observation for at least two hours after administration during the first six weeks of drug administration. Administration of the mafosfamide and sampling of the cerebrospinal fluid from the Ommaya reservoir, lumbar reservoir, or spinal tap takes about 30 minutes. In addition, after mafosfamide has been given by lumbar puncture, patients must remain lying down on their stomach for one hour.

In patients who have Ommaya reservoirs or lumbar catheters, samples of spinal fluid will be taken from the reservoirs following the first two doses of mafosfamide. For each series of tests, a total of eight spinal fluid samples will be taken with a needle from the Ommaya reservoir over a period of 24 hours after the dose. A spinal tap will be also be performed two hours after the dose on these two days. If you have a lumbar reservoir, eight spinal fluid samples will be taken with a needle from the Ommaya reservoir, over a period of 24 hours after the dose. These samples of cerebrospinal fluid will be used to measure the amount of mafosfamide found in the cerebrospinal fluid at the time they are drawn. This will help us understand how the body handles mafosfamide.

For patients with leukemia, a bone marrow aspiration (taking some bone marrow out of the pelvis bone) is necessary before receiving intrathecal mafosfamide. This is to make sure that there is no cancer in the bone marrow.

ELIGIBILITY:
* Over 3 years of age with meningeal malignancies that are progressive or refractory to conventional therapy. Patients with meningeal malignancies secondary to an underlying solid tumor are eligible at initial diagnosis if there is no conventional therapy.
* Patients with leukemia, lymphoma, or other solid tumor who also have overt meningeal involvement by their tumor.
* Must have a life expectancy of at least 8 weeks and an ECOG performance status of 2 or better.
* Must sign an informed consent indicating that they are aware of the investigational nature of this study.
* Patients must have recovered from the acute toxic effects of all prior intrathecal chemotherapy, immunotherapy, or radiotherapy, prior to entering this study and must be without significant systemic illness (e.g. infection). Patients must not have received any CNS therapy within 1 week prior to starting treatment on this study or craniospinal irradiation within 8 weeks prior to starting treatment on this study. Patients must not have received intrathecal chemotherapy within 1 week (2 weeks if prior DTC101).
* Must not have clinically significant abnormalities with regard to liver function, renal function or metabolic parameters (electrolytes, calcium and phosphorus).
* Durable Power of Attorney (DPA): A DPA must be offered to all patients ≥ 18 years of age.

Exclusion Criteria:

* Receiving other therapy (either intrathecal or systemic) designed specifically to treat their meningeal malignancy are not eligible for this study. However, patients receiving concomitant chemotherapy to control systemic or bulk CNS disease will be eligible, provided the systemic chemotherapy is not a phase I agent, an agent which significantly penetrates the CNS (e.g., high dose methotrexate, (> 1 gm/m2), thiotepa, high dose cytarabine, (> 2 gm/m2 per day), 5-fluorouracil, intravenous 6-mercaptopurine or topotecan), or an agent known to have serious unpredictable CNS side effects.
* Clinical evidence of obstructive hydrocephalus or compartmentalization of the CSF flow as documented by a radioisotope Indium111 or Technitium99-DTPA flow study are not eligible for this protocol. If a CSF flow block or compartmentalization is demonstrated, focal radiotherapy to the site of block to restore flow and a repeat CSF flow study showing clearing of the blockage is required for the patient to be eligible for the study.
* Patients who have leukemia or lymphoma and a concomitant bone marrow relapse.
* Women of childbearing age must not be pregnant or lactating.
* Patients must not have received any other systemic investigational agent within 14 days prior to, or during, study treatment. The 14 day period should be extended if the patient received any investigational agent which is known to have delayed toxicities after 14 days. Patients must not have received any other intrathecal investigational within 7 days prior to, or during, study treatment. The 7 day period should be extended if the patient received any investigational agent which is known to have delayed toxicities after 7 days or a prolonged half-life.

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 65
Dates: Start 1990-06; Study Completion 2005-09

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Children'sHospital Los Angeles, Los Angeles, California
  - Children's Hospital National Medical Center, Washington D.C., District of Columbia
  - Mayo Clinic, Jacksonville, Florida
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Pediatric Branch, National Cancer Institute, Bethesda, Maryland
  - Mayo Clinic, Rochester, Minnesota
  - M.D. Anderson Cancer Center, Houston, Texas
  - Texas Children's Hospital, Houston, Texas
  - Neurological Research Center, Bennington, Vermont
  - Children's Hospital and Medical Center, Seattle, Washington